CLINICAL TRIAL: NCT04038281
Title: The Effects of Genetic Variation in the Bitter and Fat Taste Receptor Genes on Taste Perception, Dietary Behaviour and Obesity Status
Brief Title: Genetics of Bitter and Fat Taste
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St Mary's University College (Other)
Collaborators: Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Kim Wright, Research Administrator, St Mary's University College
Other Study IDs: SMEC_2018-19_048
Record Dates: First submitted 2019-07-18; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Genetics; Taste, Altered; Diet Habit; Obesity
MeSH Terms: conditions — Dysgeusia; Feeding Behavior; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 2 ml saliva sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sensory tests — Fat, bitter taste sensitivity and food preference measurement

SUMMARY:
Obesity is an increasing problem for adults in the UK. Diets high in fat and sugar are the major contributors to weight gain. Individual differences in taste perception are a crucial factor in determining the investigator's choice of foods and an individual's sensitivity to the either bitter or fat taste compounds has been linked to a preference for different foods including sweet and high fat foods. Previous research has not comprehensively explored the effect of both fat and bitter taste sensitivity on dietary intake and obesity status. Therefore, the aim of this study is to explore the associations between genetics, fat and bitter taste sensitivity, food preference, dietary intake and obesity measures in the adult UK population.

DETAILED DESCRIPTION:
Demographic data Participants will complete a questionnaire asking about their demographics provided in Appendix. The answers to these questions will be used to control for potential confounding effects in statistical analysis.

Genetic Analysis Saliva samples (2 ml) will be collected for DNA analyses (Genefix, Isohelix, Kent, UK) and stored in the fridge at 4 °C in M201 lab at St Mary's University. DNA extraction will be carried out through use of a PSP® SalivaGene 17 DNA Kit 1011 following the standard manufacturer protocol. DNA quantification and quality control will be assessed with spectroscopy. Following this, genotyping will be carried out using prepared TaqMan® SNP genotyping assays for genes coding for bitter and fat taste receptors and a StepOnePlus thermocycler. All samples will be analysed in duplicate in accordance with the manufacturer's protocol. All genetic analyses will be carried out at St Mary's University, Twickenham.

Anthropometrics Height (m), weight (kg) and waist circumference (cm) will be recorded by the researcher team. BMI will be calculated using the equation: weight (kg)/ height (m2) ± standard deviation and waist circumference and distribution will be compared to the UK standards.

Fat and bitter taste sensitivity The Oral Fatty Acid Threshold Assessment and Ascending Forced Choice Triangle Procedure will be used to determine each participant's oleic acid (C18:1) detection threshold (fat taste sensitivity). Briefly, each participant will be presented with three cups containing 30 ml vehicles in a random arrangement, two controls and the third containing oleic acid (0.02, 0.06, 1, 1.4, 2, 2.8, 3.8, 5, 6.4, 8, 9.8, 12, 20 mM). Participants will have to identify the oleic acid solution by tasting but not ingesting the solutions. A participant will be required to choose the oleic acid solution correctly three times at the same concentration to define their threshold. If participant is incorrect at any point, further three cups will be presented, one containing the higher concentration. There will be thirteen concentrations in total. The bitter taste compound used to classify participants into bitter taste hypo-, normal- and hypertasters will be PTC. Participants will place a strip on the tongue and use the general Labeled Magnitude Scale (gLMS) to report the intensity of the taste compound.

Food preference Food preference will be measured by asking participants to taste food usually perceived as bitter (dark chocolate and broccoli) as well as food that are defined as sweet (milk chocolate and carrots).To minimise variability, the vegetables will be presented raw. Overall preference will be tested using a nine-point Likert scale. Each participants will rinse their mouth with water between each food and a minimum of one minute will be left between each test. Eating behaviour will be determined by use of the validated Adult Eating Behaviour Questionnaire. Fat preference will be determined by a UK adaption of the validated Fat Preference Questionnaire.

Dietary Intake The validated EPIC Norfolk Food Frequency Questionnaire (FFQ) will be used to measure dietary intake over the previous year.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults aged 18-65 years

Exclusion Criteria:

* pregnancy
* breastfeeding
* smoking
* reported any past or present food allergy or lactose intolerance
* under any medication that might affect taste perception
* known illnesses such as cold, ear infection, sinus infection, or flu
* any reported chronic diseases such as (diabetes, CVD, stroke, epilepsy, asthma, cancer)
* any thyroid problems
* individuals that are currently following a diet or weight loss programme

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Caucasian males and females aged 18-65 years
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-15 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Obesity | 1 day observation
  BMI

SECONDARY OUTCOMES:
Energy intake | 1 year dietary intake
  Energy intake in kcal obtained with FFQ
Fat intake | 1 year dietary intake
  Fat intake in grams obtained with FFQ
Sugar intake | 1 year dietary intake
  Sugar intake in grams obtained with FFQ

CONTACTS AND LOCATIONS:
Locations (1):
- St Mary's University, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No